CLINICAL TRIAL: NCT05669261
Title: A PILOT STUDY ON RESEARCH TREATMENT OF LONG COVID POST-ACUTE SEQUELAE OF SARS CoV-2 INFECTION ("PASC") USING ATCell™
Brief Title: Treatment of Long COVID Symptoms Utilizing Autologous Stem Cells Following COVID-19 Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American CryoStem Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0001_CRYO_LC19_ADSC_001
Record Dates: First submitted 2022-12-21; First posted 2022-12-30 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Long COVID
Keywords: Long COVID; Post Acute Sequelae
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Lipectomy

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized single-center, double-blinded, placebo controlled standard of care plus study. Once safety has been certified by IRB/ HRPP, the study will be unblinded and participants that received the placebo treatment will be offered the opportunity to crossover and receive 150 million cell ATCell™ autologous treatment with the same monitoring and clinical support afforded to the first treatment cohort
Who Masked: Participant, Care Provider, Investigator
Masking Description: To ensure proper Randomization, the Sponsor has elected to use the NIH National Cancer Institute Clinical Trial Randomization tool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATCell Treatment Group (Experimental): A single administration of expanded autologous lines at a total dose exposure of 150 million cells ("ATCell™") will be administered to this group.
  Interventions: Procedure: Adipose Tissue Harvest; Biological: ATCell
- Placebo (Placebo Comparator): a single administration of Placebo (Sham Treatment) IV infusion of Ringers Lactate with 5% Dextrose will be administered to this group.
  Interventions: Procedure: Adipose Tissue Harvest

INTERVENTIONS:
Procedure: Adipose Tissue Harvest — Local Anesthesia will be administered. A Stab wound will be created at the harvest site through which a 3.0 or 2.5 mm cannula will be inserted to suction fat using the "syringe" (i.e. manual) technique. A total of 100 cc of lipoaspirate will be collected by manual draw of the adipose tissue into syringes.
  Other Names: Liposuction
Biological: ATCell — Infusion of the study medication at the rate of 575 mL/HR (500ml of LRD5 plus 75ml of ATCell suspended in LRD5) and continue until all received trial medication has been delivered.
  Other Names: Autologous Adipose Derived Mesenchymal Stem Cells
  Arms: ATCell Treatment Group

SUMMARY:
The project is described as a Phase 1 Clinical Safety Study intended to provide preliminary assessments of the safety, tolerability, and secondarily to be vigilant for signals of amelioration of symptoms associated with Post-Acute Sequelae of SARS-CoV-2 infection

DETAILED DESCRIPTION:
The proposed study is a randomized single-center, double-blinded, placebo controlled standard of care plus study. Each participant will continue to receive standard of care treatment for their current diagnosis and be afforded the opportunity to add any additional care as needed that may include care for behavioral health concerns. In the proposed study, safety of a single administration of expanded autologous lines at a total dose exposure of 150 million cells ("ATCell™") will be assessed. Each ATCell™ cell batch will be derived from ex vivo expanded stromal vascular fraction (SVF) of a participant's own adipose tissue. SVF is collected by liposuction and expanded. Briefly, ATCell suspended in Lactated Ringer's with 5% dextrose solution, or a placebo of Lactated Ringers 5% dextrose solution will be administered once to each participant. Safety will be evaluated through clinical assessments and laboratory test results comparing treatment cohort participant's baseline assessments and laboratory test results. Following completion of follow up period as defined in the schedule of events, the study will be unblinded, the results reviewed by the Institutional Review Board (IRB) and Human Research Protection Program (HRPP). Once safety has been reviewed by IRB/ HRPP, the study will be unblinded and participants that received the placebo treatment will be offered the opportunity to crossover and receive 150 million cell ATCell™ autologous treatment with the same monitoring and clinical support afforded to the first treatment cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty service members: military retirees, DEERS eligible dependents who are Tricare beneficiaries only (Department of Defense (DoD) investigational sites only)
2. Participants ages of 18 years and above
3. Documentation of a positive COVID-19 polymerase chain reaction (PCR) test or strong history of SARS-CoV-2 exposure with positive supportive serology
4. Male or female or other gender
5. Individuals with established diagnosis of PASC
6. Subjects with moderate to severe levels of PASC based on synthesis of multiple assessment modalities provided by the multispecialty study team.
7. PASC phenotype to include signs and symptoms of fatigue and low endurance and either Autonomic Disorder or Dyspnea or both.
8. Subjects who are able to comprehend the consent procedure and follow the treatment process.
9. Female participants of childbearing potential and at risk of pregnancy during the study must agree to use 2 highly effective methods of contraception throughout the study and for 112 days after the last study visit.
10. Female participant who are not of childbearing potential (i.e,. must meet at least one (1) of the following criteria): have undergone a hysterectomy and/or bilateral oophorectomy, or ovarian failure .
11. For male subjects who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception, willingness to use a barrier method of contraception (condom) from the start of study therapy until ≥ 90 days after the end of the study and to refrain from sperm donation until ≥ 90 days after the end of the study.
12. Achieved postmenopausal status defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or psychological cause and have a serum follicle stimulating hormone (FSH) level confirming the post-menopausal state.
13. Individuals who are willing and able to comply with lifestyle guidelines, scheduled visits, treatment plan, laboratory tests, and other study procedures through the end of the final study visit.
14. Individuals with the following Vital Signs:

    1. Systolic Blood Pressure of > 100 or < 140 (mmHg)
    2. Diastolic Blood Pressure of > 60 or <90 (mmHg)
    3. Heart Rate of > 60 or < 100 (bpm) (beats per minute)
    4. Temperature of < 38°C (afebrile)
    5. Respiratory Rate of > 12 or < 20 (bpm) (breaths per minute)
    6. Pulse Ox greater than >95% on room air
    7. BMI < 28

Exclusion Criteria:

5.3.7.4 Exclusion Criteria:

1. Subjects with documented past or current history of severe depression, suicidal ideations or suicidal attempts.
2. Subjects who are unable to comprehend the content of informed consent
3. Female subjects who are pregnant or who are not willing to practice effective contraception during and for 112 days following the last study visit
4. Female subjects who are breastfeeding
5. History of abnormal brain or spinal MRI for presence of thromboembolic events.
6. Recent traumatic brain injury or other concussive event within 12 months of medical history review
7. History of abnormal Echocardiogram for cardiac structure or function in the last 10 years.
8. Prior history of postural orthostatic tachycardia syndrome predating diagnosis of SARS-CoV2 infection
9. Uncontrolled hypertension or hyperlipidemia
10. Prior to COVID diagnosis, the presence of abnormal chest x-ray for any parenchymal disease, or,

    1. Active tuberculosis or ongoing treatment for tuberculosis or any acute or chronic infection affecting lung
    2. Chronic lung disease due to fibrosis or autoimmune inflammation such as sarcoidosis or rheumatoid arthritis, vasculitis or lupus
    3. Lung cancer
    4. Asthma
    5. Chronic obstructive pulmonary disease (COPD)
    6. Emphysema
    7. Disorders of upper airway, larynx, or trachea that pose potential complications in a state of emergency for airway management due to SAE.
    8. Disorders of pleura that affects pulmonary functions
11. Prior history of connective tissue diseases
12. History of severe hospitalization from COVID-19 or other respiratory infection requiring mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
13. Pulse oxygenation readings <95% on room air during screening exam
14. History of pulmonary embolism during lifetime
15. Prior history of deep venous thromboses, stroke or myocardial infarction
16. Any thrombophilia, including factor V Leiden, protein C deficiency, and protein S deficiency
17. Ongoing pharmaceutical or radiation treatment for infection or malignancy
18. Prior positive test for any of the following without demonstration of resolution: viral Hepatitis B or C (HBV, HCV), Human Immunodeficiency virus -1 or -2 (HIV1 or HIV2), Human T cell leukemia virus -I or -II (HTLV-1 or HTLV-II), West Nile, Zika, Syphilis.
19. Use of any immunosuppressive, immune modulating drugs include calcineurin inhibitors, antimetabolites, alkylating agents, for greater than 14 consecutive days over the last 3 months
20. Actively listing (or expected listing) for transplant of any organ, other than corneal, bone, skin, ligament or tendon transplant.
21. Be an organ transplant recipient in the past, other than for corneal, bone, skin, ligament or tendon transplant.
22. History of malignant tumor within the past 10 years for breast cancer and 5 years for all other cancers.
23. Individuals allergic to local anesthetics
24. Individuals with inadequate subcutaneous tissue to allow appropriate lipoaspirate (i.e., fat extraction)
25. Any history of autoimmune illnesses including but not limited to: Multiple sclerosis, Crohn's disease, Myasthenia gravis, Hashimoto's thyroiditis, psoriatic arthritis, Pernicious anemia/atrophic gastritis, Guillain-Barre, Chronic inflammatory demyelinating polyneuropathy, Type 1 diabetes mellitus, Inflammatory bowel disease, Systemic lupus erythematosus, vasculitis, Immune thrombocytopenic purpura, inflammatory muscle disease or Rheumatoid arthritis, Rheumatic fever.
26. Uncontrolled type 2 diabetes
27. Any abnormal test result, in the opinion of the PI and the study team, that may compromise the safety or compliance of the participant or preclude successful completion of the study, or that may compromise the validity of the study.
28. Individuals expecting retirement, military separation, deployment or relocation in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Incidence of Serious Adverse Events (SAEs) | Upon completion of final post treatment clinical visit of all participants
  Observed Adverse Events (AE's) in the placebo control group will be compared to observed AE in the experimental treatment, if any, in order to assess safety of the experimental treatment.
Assessment of change in Health Status using the 36 item Short Form Health Survey (SF-36) | One week post administration
  Completed by Participant as a part of physician visits at baseline, and once per week following treatment. Scores of completed SF-36 will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative).The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Assessment of change in Health Status using the 36 item Short Form Health Survey (SF-36) | Two weeks post administration
  Completed by Participant as a part of physician visits at baseline, and once per week following treatment. Scores of completed SF-36 will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative).The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Assessment of change in Health Status using the 36 item Short Form Health Survey (SF-36) | Three weeks post administration
  Completed by Participant as a part of physician visits at baseline, and once per week following treatment. Scores of completed SF-36 will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative).The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Assessment of change in Health Status using the 36 item Short Form Health Survey (SF-36) | Four weeks post administration
  Completed by Participant as a part of physician visits at baseline, and once per week following treatment. Scores of completed SF-36 will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative).The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

SECONDARY OUTCOMES:
Assessment of Changes in Exosome/Cytokine/Chemokine Testing | Once per week for four weeks post administration
  Blood samples will be collected for testing to measure the selected cytokine and chemokines blood panels described below at screening (baseline), at the pre-treatment clinical visit, and the one- and four-week clinical visits following treatment
Assessment of change in completion time -Six-minute walk test (6MWT) | Four weeks post administration
  The 6MWT is a self-paced walking test in which the subject is instructed to walk as fast as possible for 6 minutes. The 6WMT will be completed by each participant at the screening, pre-Treatment clinical visit and at the one week and four week post treatment clinical visits.
Assessment of Change in Complete blood count with differential (CBC with diff) Laboratory Testing Results | Each week for four weeks post administration
  Complete blood count with differential (CBC with diff)Test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline
Assessment of Change in Lactate dehydrogenase (LDH) Laboratory Testing Results | Each week for four weeks post administration
  Lactate dehydrogenase (LDH) test results are to be assessed in this study are complete blood count with differential (CBC with diff), to identify any significant change in results positive or negative with the change reported as a percentage change from baseline
Assessment of Change in Prothrombin time/partial thromboplastin time (PT/PTT Coagulation factors II) Laboratory Testing Results | Each week for four weeks post administration
  Prothrombin time/partial thromboplastin time (PT/PTT Coagulation factors II) test results are to be assessed to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.
Assessment of Change in Troponin Laboratory Testing Results | Each week for four weeks post administration
  Troponin test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.
Assessment of Change in D-dimer Laboratory Testing Results | Each week for four weeks post administration
  D-dimer test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.
Assessment of Change in Fibrinogen (Coagulation factors II) Laboratory Testing Results | Each week for four weeks post administration
  Fibrinogen (Coagulation factors II) test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.
Assessment of Change in estimated glomerular filtration rate Laboratory Testing Results | Each week for four weeks post administration
  estimated glomerular filtration rate (eGFR) test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.
Assessment of Change in Urinalyses Laboratory Testing Results | Each week for four weeks post administration
  Urinalyses test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.
Assessment of Change in Spot creatinine Laboratory Testing Results | Each week for four weeks post administration
  Spot creatinine test results are to be assessed in this study to identify any significant change in results positive or negative with the change reported as a percentage change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Y Dudzinski, Study Director — American CryoStem Corporation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nasserie T, Hittle M, Goodman SN. Assessment of the Frequency and Variety of Persistent Symptoms Among Patients With COVID-19: A Systematic Review. JAMA Netw Open. 2021 May 3;4(5):e2111417. doi: 10.1001/jamanetworkopen.2021.11417. PMID 34037731
- [Background] Alkodaymi MS, Omrani OA, Ashraf N, Shaar BA, Almamlouk R, Riaz M, Obeidat M, Obeidat Y, Gerberi D, Taha RM, Kashour Z, Kashour T, Berbari EF, Alkattan K, Tleyjeh IM. Prevalence of post-acute COVID-19 syndrome symptoms at different follow-up periods: a systematic review and meta-analysis. Clin Microbiol Infect. 2022 May;28(5):657-666. doi: 10.1016/j.cmi.2022.01.014. Epub 2022 Feb 3. PMID 35124265
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Nehme M, Braillard O, Alcoba G, Aebischer Perone S, Courvoisier D, Chappuis F, Guessous I; COVICARE TEAM. COVID-19 Symptoms: Longitudinal Evolution and Persistence in Outpatient Settings. Ann Intern Med. 2021 May;174(5):723-725. doi: 10.7326/M20-5926. Epub 2020 Dec 8. No abstract available. PMID 33284676
- [Background] Garrigues E, Janvier P, Kherabi Y, Le Bot A, Hamon A, Gouze H, Doucet L, Berkani S, Oliosi E, Mallart E, Corre F, Zarrouk V, Moyer JD, Galy A, Honsel V, Fantin B, Nguyen Y. Post-discharge persistent symptoms and health-related quality of life after hospitalization for COVID-19. J Infect. 2020 Dec;81(6):e4-e6. doi: 10.1016/j.jinf.2020.08.029. Epub 2020 Aug 25. PMID 32853602
- [Background] Ladds E, Rushforth A, Wieringa S, Taylor S, Rayner C, Husain L, Greenhalgh T. Persistent symptoms after Covid-19: qualitative study of 114 "long Covid" patients and draft quality principles for services. BMC Health Serv Res. 2020 Dec 20;20(1):1144. doi: 10.1186/s12913-020-06001-y. PMID 33342437
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Jin Y, Ji W, Yang H, Chen S, Zhang W, Duan G. Endothelial activation and dysfunction in COVID-19: from basic mechanisms to potential therapeutic approaches. Signal Transduct Target Ther. 2020 Dec 24;5(1):293. doi: 10.1038/s41392-020-00454-7. PMID 33361764
- [Background] Bocci M, Oudenaarden C, Saenz-Sarda X, Simren J, Eden A, Sjolund J, Moller C, Gisslen M, Zetterberg H, Englund E, Pietras K. Infection of Brain Pericytes Underlying Neuropathology of COVID-19 Patients. Int J Mol Sci. 2021 Oct 27;22(21):11622. doi: 10.3390/ijms222111622. PMID 34769052
- [Background] Cardot-Leccia N, Hubiche T, Dellamonica J, Burel-Vandenbos F, Passeron T. Pericyte alteration sheds light on micro-vasculopathy in COVID-19 infection. Intensive Care Med. 2020 Sep;46(9):1777-1778. doi: 10.1007/s00134-020-06147-7. Epub 2020 Jun 12. No abstract available. PMID 32533198
- [Background] Jones OY, Yeralan S. Is Long COVID a State of Systemic Pericyte Disarray? J Clin Med. 2022 Jan 24;11(3):572. doi: 10.3390/jcm11030572. PMID 35160024
- [Background] Munir H, McGettrick HM. Mesenchymal Stem Cell Therapy for Autoimmune Disease: Risks and Rewards. Stem Cells Dev. 2015 Sep 15;24(18):2091-100. doi: 10.1089/scd.2015.0008. Epub 2015 Jul 28. PMID 26068030
- [Background] Mezey E, Nemeth K. Mesenchymal stem cells and infectious diseases: Smarter than drugs. Immunol Lett. 2015 Dec;168(2):208-14. doi: 10.1016/j.imlet.2015.05.020. Epub 2015 Jun 4. PMID 26051681
- [Background] Arabpour E, Khoshdel S, Tabatabaie N, Akhgarzad A, Zangiabadian M, Nasiri MJ. Stem Cells Therapy for COVID-19: A Systematic Review and Meta-Analysis. Front Med (Lausanne). 2021 Nov 29;8:737590. doi: 10.3389/fmed.2021.737590. eCollection 2021. PMID 34912818
- [Background] Golchin A, Seyedjafari E, Ardeshirylajimi A. Mesenchymal Stem Cell Therapy for COVID-19: Present or Future. Stem Cell Rev Rep. 2020 Jun;16(3):427-433. doi: 10.1007/s12015-020-09973-w. PMID 32281052
- [Background] Worm-Smeitink M, Gielissen M, Bloot L, van Laarhoven HWM, van Engelen BGM, van Riel P, Bleijenberg G, Nikolaus S, Knoop H. The assessment of fatigue: Psychometric qualities and norms for the Checklist individual strength. J Psychosom Res. 2017 Jul;98:40-46. doi: 10.1016/j.jpsychores.2017.05.007. Epub 2017 May 8. PMID 28554371
- [Background] Plash WB, Diedrich A, Biaggioni I, Garland EM, Paranjape SY, Black BK, Dupont WD, Raj SR. Diagnosing postural tachycardia syndrome: comparison of tilt testing compared with standing haemodynamics. Clin Sci (Lond). 2013 Jan;124(2):109-14. doi: 10.1042/CS20120276. PMID 22931296